CLINICAL TRIAL: NCT07167459
Title: A Phase II Trial of Personalized Definitive Stereotactic Body Radiotherapy (SBRT) for Early-Stage Peripheral Non-Small Cell Lung Cancer (NSCLC) With Correlative Omics Analysis
Brief Title: Personalized SBRT in Early-Stage Peripheral NSCLC
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20230372; TZ3582022-005 (Other Grant/Funding Number: Tianjin Medical University Cancer Institute and Hospital)
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Early-stage Peripheral Non-small Cell Lung Cancer
MeSH Terms: interventions — Radiosurgery; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized SBRT for Early-Stage Peripheral NSCLC (Experimental): This single-arm cohort comprises patients with newly diagnosed, early-stage peripheral non-small-cell lung cancer (T1-2N0M0, IA-IIA) who receive individualized stereotactic body radiotherapy (SBRT) as standard-of-care. Participants will be prospectively followed for 3 years to assess overall survival, local control, progression-free survival, and adverse events. Inclusion criteria: age ≥18 years, pathologically confirmed NSCLC, tumor location ≥2 cm from the proximal bronchial tree, ECOG 0-2, and medically inoperable or refusal of surgery.
  Interventions: Device: ndividualized Stereotactic Body Radiotherapy (SBRT) System

INTERVENTIONS:
Device: ndividualized Stereotactic Body Radiotherapy (SBRT) System — The individualized SBRT system employs advanced image-guided radiation delivery to deliver highly conformal, ablative doses to early-stage peripheral non-small-cell lung cancer while minimizing exposure to surrounding normal tissues. Treatment is delivered via a state-of-the-art robotic radiosurgery platform (e.g., CyberKnife M6) according to patient-specific fractionation schedules based on tumor size and proximity to critical structures, following standard indications and institutional protocols for medically inoperable or surgically refused cases.

SUMMARY:
This study aims to learn about the long-term safety and effectiveness of personalized stereotactic body radiotherapy (SBRT) in patients with early-stage peripheral non-small cell lung cancer (NSCLC). Individualized SBRT is a specialized radiation technique that delivers precise, high-dose treatment while minimizing damage to surrounding normal tissues.

The main question it aims to answer is:

Does individualized SBRT maintain local tumor control and patient survival at 3 years without significant side effects?

Patients with early-stage peripheral NSCLC who are medically inoperable or refuse surgery, and who are scheduled to receive individualized SBRT as their standard treatment, will provide the data to assess the safety and efficacy of this personalized radiation approach.

ELIGIBILITY:
Inclusion Criteria

* Participant or legal guardian provides written informed consent.
* Age ≥18 years; no upper age limit; male or female.
* Pathologically confirmed non-small-cell lung cancer (NSCLC) staged T1-2N0M0 (IA-IIA, AJCC 8th ed.).
* Peripheral tumor location: ≥2 cm from the proximal bronchial tree or any mediastinal structure.
* Medically inoperable (e.g., FEV1 <40 % predicted, DLCO <40 % predicted, NYHA class III-IV heart failure) or refusal of surgery.
* ECOG performance status 0-2.
* Life expectancy ≥6 months per investigator judgment.
* Measurable disease by RECIST 1.1.
* Adequate organ function (blood counts, liver and renal indices) per institutional standards.
* Willing and able to comply with all study procedures, imaging schedules, and follow-up visits.
* Effective contraception for women of child-bearing potential and fertile men for 12 months after SBRT completion.

Exclusion Criteria

* Previous thoracic radiotherapy, chemotherapy, targeted therapy, or surgery for lung cancer.
* Evidence of regional or distant metastases.
* Concurrent or prior malignancy within 5 years (except adequately treated basal-cell carcinoma of skin or carcinoma in situ of cervix).
* Active interstitial pneumonitis, radiation pneumonitis, drug-induced pneumonitis, or clinically significant pulmonary fibrosis.
* Pregnancy, lactation, or planned pregnancy.
* Participation in another interventional clinical trial with an unmet primary endpoint.
* Known psychiatric disorder, substance abuse, or other condition that would impair compliance.
* Contraindication to contrast-enhanced CT or PET-CT imaging.
* Investigator-determined medical, social, or psychological contraindications that could compromise safety or data integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival (OS) | Approximately 36 months after enrollment
  Three-year overall survival is defined as the proportion of participants who remain alive at 36 months from the start of individualized stereotactic body radiotherapy (SBRT).

SECONDARY OUTCOMES:
3-year Progression-Free Survival (PFS) | Enrollment → 36 months
  Proportion of participants alive and without radiographic progression at 36 months.
3-year Local Control (LC) | Enrollment → 36 months
  Proportion of participants with no evidence of tumor recurrence at the irradiated site at 36 months.
Objective Response Rate (ORR) | Enrollment → ~5 months (≈1 month to complete SBRT plus 4 months follow-up)
  Percentage of participants achieving complete or partial response per RECIST 1.1 at 4 months after SBRT completion.
Adverse Event Incidence | Enrollment → 6 months after last SBRT fraction
  Frequency and severity of all treatment-related toxicities graded by CTCAE 5.0, collected continuously.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin Key Laboratory of Cancer Prevention and Therapy, Tianjin, Tianjin 300060, Tianjin, Tianjin Municipality, China